CLINICAL TRIAL: NCT01938378
Title: An Open-label, Multicenter, Post-Marketing Requirement Study to Investigate the Safety and Tolerability of Octaplas™ in the Management of Pediatric Patients Who Require Therapeutic Plasma Exchange
Brief Title: Octaplas Pediatric Plasma Exchange Trial
Acronym: Octaplas
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAS-213
Record Dates: First submitted 2013-09-02; First posted 2013-09-10 (Estimated); Results first posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Adverse Effects in the Therapeutic Use of Plasma Substitutes
Keywords: Octaplas

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pediatric patients undergoing TPE (Other): octaplas™
  Interventions: Biological: Octaplas™

INTERVENTIONS:
Biological: Octaplas™ — octaplas™ infusion solution for IV administration, ABO compatibile. Recommended dose for a plasma exchange is 40 to 60 ml/kg.
  Other Names: octaplas

SUMMARY:
To assess the safety and tolerability of octaplas™ in the pediatric population by monitoring serious adverse drug reactions, adverse drug reactions (ADRs), thrombotic events (TEs), thromboembolic events (TEEs) and by measuring safety laboratory parameters in pediatric patients who require therapeutic plasma exchange.

ELIGIBILITY:
Inclusion Criteria:

1. Patients in whom therapeutic plasma exchange (TPE) is required.
2. Patient is male or female ≥ 2 years to ≤ 20 years of age.
3. Patient or patient's legal representative(s)/guardian(s) has /have given voluntarily written and signed informed consent before any study-related procedure is to be performed. If children are old enough (age usually deemed by each institution) to understand the risks and benefits of the study, they should also be informed and provide their written assent.

Exclusion Criteria:

1. Patient with known homozygous congenital deficiency of Protein S.

   Exclusion Criteria:
2. Patient has a history of severe hypersensitivity reaction to plasma-derived products or to any excipient of the investigational product.
3. Patient has an already known IgA deficiency with documented antibodies against IgA.
4. Patient is currently participating in another interventional clinical study or has participated during the past 1 month prior to study inclusion. This is not applicable to non-interventional trials and does not exclude patients who have been exposed to Investigational Medicinal Product with a washout of at least 30 days from enrollment in LAS-213. Concurrent participation in a device study will be considered on a case by case basis.
5. Patient is pregnant.
6. Use of Angiotensin-Converting-Enzyme-inhibitors within 72 hours of the start of the first infusion episode or planned used of these medications while on study.

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2015-04; Primary Completion 2019-01-27 (Actual); Study Completion 2019-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Frenzel, MD, Study Director — Medical Director
Locations (8):
- United States (8):
  - Octapharma Research Site, Birmingham, Alabama
  - Octapharma Research Site, Atlanta, Georgia
  - Octapharma Research Site, New Orleans, Louisiana
  - Octapharma Research Site, Minneapolis, Minnesota
  - Octapharma Research Site, Kansas City, Missouri
  - Octapharma Research Site, St Louis, Missouri
  - Octapharma Research Site, Durham, North Carolina
  - Octapharma Research Site, Cincinnati, Ohio

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pediatric Patients Undergoing TPE
Started | 41
Completed | 41
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Pediatric Patients Undergoing TPE Age Group 1: Ages 2-<12
- Pediatric Patients Undergoing TPE Age Group 2: Ages 12-<17
- Pediatric Patients Undergoing TPE Age Group 3: Ages ≥17
- Total: Total of all reporting groups
Arm/Group | Pediatric Patients Undergoing TPE Age Group 1 | Pediatric Patients Undergoing TPE Age Group 2 | Pediatric Patients Undergoing TPE Age Group 3 | Total
Number analyzed (Participants) | 15 | 13 | 13 | 41
Age, Continuous [Median (Standard Deviation); unit: years] | 6.1 (2.34) | 13.8 (1.52) | 18.1 (1.04) | 12.3 (5.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 4 | 23
  Male | 3 | 6 | 9 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 15 | 12 | 12 | 39
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 2
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 3 | 7
  White | 13 | 9 | 10 | 32
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Monitoring of Adverse Drug Reactions Caused by the Octaplas™Used for Plasma Exchange.
Description: Monitoring of adverse drug reactions caused by the octaplas™used for plasma exchange.
Time Frame: up to 8 days including the 24 hour follow-up from treatment
Measure: Number; unit: event
Groups:
- Pediatric Patients Undergoing TPE Age Group 2: Ages 12 - <17
- All Patients: All ages
Arm/Group | Pediatric Patients Undergoing TPE Age Group 1 | Pediatric Patients Undergoing TPE Age Group 2 | Pediatric Patients Undergoing TPE Age Group 3 | All Patients
Number analyzed (Participants) | 15 | 13 | 13 | 41
event | 0 | 5 | 3 | 8

2. Primary Outcome: Monitoring of TEs and TEEs Caused by the Octaplas™Used for Plasma Exchange.
Description: Monitoring of Thrombotic Events (TEs) and Thromboembolic Events (TEEs) caused by the octaplas™used for plasma exchange.
Time Frame: up to 8 days including the 24 hour follow-up from treatment
Measure: Number; unit: event
Arm/Group | Pediatric Patients Undergoing TPE Age Group 1 | Pediatric Patients Undergoing TPE Age Group 2 | Pediatric Patients Undergoing TPE Age Group 3 | All Patients
Number analyzed (Participants) | 15 | 13 | 13 | 41
event | 0 | 0 | 0 | 0

3. Secondary Outcome: Assessment of Blood Urea Nitrogen Levels
Description: Blood samples compare levels before each TPE (therapeutic plasma exchange) and after each TPE. Pre-TPE is within 24 hours before TPE start; Post-TPE is 30 minutes to 3 hours after TPE end.
Time Frame: up to 8 days including the 24 hour follow-up
Population: Not all patients received blood draws/multiple TPEs
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Pre-TPE: Value pre-TPE
- Post-TPE: Value post-TPE
- Change From Pre-TPE: Change in level from Pre-TPE to Post-TPE
Arm/Group | Pre-TPE | Post-TPE | Change From Pre-TPE
Number analyzed (Participants) | 41 | 41 | 41
mg/dL
  TPE 1: number analyzed (Participants) | 39 | 36 | 34
  TPE 1 | 26.4 (18.69) | 25.2 (18.22) | -1.4 (6.56)
  TPE 2: number analyzed (Participants) | 24 | 18 | 17
  TPE 2 | 27.3 (19.31) | 27.6 (18.67) | 1.2 (4.69)
  TPE 3: number analyzed (Participants) | 18 | 11 | 11
  TPE 3 | 32.5 (25.47) | 26.4 (25.29) | 1.1 (3.21)
  TPE 4: number analyzed (Participants) | 10 | 8 | 8
  TPE 4 | 28.3 (14.38) | 28.6 (16.21) | 1.5 (2.67)
  TPE 5: number analyzed (Participants) | 6 | 4 | 4
  TPE 5 | 31.2 (18.95) | 35.5 (25.12) | -0.5 (4.36)
  TPE 6: number analyzed (Participants) | 1 | 1 | 1
  TPE 6 | 21.0 (0) | 20.0 (0) | -1.0 (0)

4. Secondary Outcome: Assessment of Carbon Dioxide Levels
Description: as for outcome 3
Time Frame: up to 8 days including the 24 hour follow-up
Population: Not all patients received blood draws/multiple TPEs
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Pre-TPE | Post-TPE | Change From Pre-TPE
Number analyzed (Participants) | 41 | 41 | 41
mmol/L
  TPE 1: number analyzed (Participants) | 39 | 36 | 34
  TPE 1 | 25.0 (4.04) | 26.9 (4.62) | 2.2 (3.03)
  TPE 2: number analyzed (Participants) | 24 | 18 | 17
  TPE 2 | 27.3 (3.58) | 28.2 (3.96) | 0.5 (2.79)
  TPE 3: number analyzed (Participants) | 18 | 11 | 11
  TPE 3 | 26.2 (3.13) | 26.7 (2.33) | 1.2 (1.72)
  TPE 4: number analyzed (Participants) | 10 | 8 | 8
  TPE 4 | 26.3 (3.13) | 26.6 (4.87) | 1.0 (2.98)
  TPE 5: number analyzed (Participants) | 6 | 4 | 4
  TPE 5 | 27.3 (4.32) | 27.0 (7.75) | 0.3 (5.50)
  TPE 6: number analyzed (Participants) | 1 | 1 | 1
  TPE 6 | 29.0 (0) | 32.0 (0) | 3.0 (0)

5. Secondary Outcome: Assessment of Chloride Levels
Description: as for outcome 3
Time Frame: up to 8 days including the 24 hour follow-up
Population: Not all patients received blood draws/multiple TPEs
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Pre-TPE | Post-TPE | Change From Pre-TPE
Number analyzed (Participants) | 41 | 41 | 41
mmol/L
  TPE 1: number analyzed (Participants) | 39 | 36 | 34
  TPE 1 | 105.0 (4.24) | 105.2 (5.15) | 0.5 (3.31)
  TPE 2: number analyzed (Participants) | 24 | 18 | 17
  TPE 2 | 105.5 (4.44) | 105.4 (5.04) | 0.6 (2.72)
  TPE 3: number analyzed (Participants) | 18 | 11 | 11
  TPE 3 | 106.7 (5.28) | 107.5 (6.15) | -0.3 (2.37)
  TPE 4: number analyzed (Participants) | 10 | 8 | 8
  TPE 4 | 106.4 (7.06) | 106.8 (6.98) | -0.9 (2.59)
  TPE 5: number analyzed (Participants) | 6 | 4 | 4
  TPE 5 | 103.0 (5.22) | 104.8 (7.93) | 1.0 (6.78)
  TPE 6: number analyzed (Participants) | 1 | 1 | 1
  TPE 6 | 111.0 (0) | 108.0 (0) | -3.0 (0)

6. Secondary Outcome: Assessment of Creatinine Levels
Description: as for outcome 3
Time Frame: up to 8 days including the 24 hour follow-up
Population: Not all patients received blood draws/multiple TPEs
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Pre-TPE | Post-TPE | Change From Pre-TPE
Number analyzed (Participants) | 41 | 41 | 41
mg/dl
  TPE 1: number analyzed (Participants) | 39 | 36 | 34
  TPE 1 | 1.7 (2.24) | 1.3 (1.45) | -0.4 (1.10)
  TPE 2: number analyzed (Participants) | 24 | 18 | 17
  TPE 2 | 1.3 (1.00) | 1.2 (0.95) | -0.1 (0.31)
  TPE 3: number analyzed (Participants) | 18 | 11 | 11
  TPE 3 | 1.1 (0.78) | 0.9 (0.84) | -0.1 (0.22)
  TPE 4: number analyzed (Participants) | 10 | 8 | 8
  TPE 4 | 1.0 (0.51) | 0.9 (0.59) | 0.0 (0.09)
  TPE 5: number analyzed (Participants) | 6 | 4 | 4
  TPE 5 | 1.1 (0.66) | 1.2 (0.87) | 0.1 (0.09)
  TPE 6: number analyzed (Participants) | 1 | 1 | 1
  TPE 6 | 0.8 (0) | 0.8 (0) | 0.0 (0.0)

7. Secondary Outcome: Assessment of Glucose Levels
Description: as for outcome 3
Time Frame: up to 8 days including the 24 hour follow-up
Population: Not all patients received blood draws/multiple TPEs
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Pre-TPE | Post-TPE | Change From Pre-TPE
Number analyzed (Participants) | 41 | 41 | 41
mg/dl
  TPE 1: number analyzed (Participants) | 39 | 36 | 34
  TPE 1 | 144.7 (70.10) | 135.2 (41.89) | -12.0 (65.83)
  TPE 2: number analyzed (Participants) | 24 | 18 | 17
  TPE 2 | 138.2 (61.92) | 142.7 (75.86) | 12.5 (44.76)
  TPE 3: number analyzed (Participants) | 18 | 11 | 11
  TPE 3 | 141.9 (65.12) | 156.9 (57.67) | 22.6 (45.69)
  TPE 4: number analyzed (Participants) | 10 | 8 | 8
  TPE 4 | 191.0 (142.81) | 142.1 (59.04) | -44.3 (158.61)
  TPE 5: number analyzed (Participants) | 6 | 4 | 4
  TPE 5 | 147.2 (85.33) | 140.8 (61.70) | 15.8 (38.59)
  TPE 6: number analyzed (Participants) | 1 | 1 | 1
  TPE 6 | 77.0 (0) | 75.0 (0) | -2.0 (0)

8. Secondary Outcome: Assessment of Potassium Levels
Description: as for outcome 3
Time Frame: up to 8 days including the 24 hour follow-up
Population: Not all patients received blood draws/multiple TPEs
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Pre-TPE | Post-TPE | Change From Pre-TPE
Number analyzed (Participants) | 41 | 41 | 41
mmol/L
  TPE 1: number analyzed (Participants) | 39 | 36 | 34
  TPE 1 | 3.9 (0.57) | 3.8 (0.58) | -0.1 (0.54)
  TPE 2: number analyzed (Participants) | 24 | 18 | 17
  TPE 2 | 3.9 (0.43) | 4.0 (0.47) | 0.1 (0.26)
  TPE 3: number analyzed (Participants) | 18 | 11 | 11
  TPE 3 | 3.7 (0.57) | 3.9 (0.36) | 0.1 (0.49)
  TPE 4: number analyzed (Participants) | 10 | 8 | 8
  TPE 4 | 4.1 (0.62) | 4.0 (0.64) | -0.2 (0.65)
  TPE 5: number analyzed (Participants) | 6 | 4 | 4
  TPE 5 | 3.9 (0.30) | 3.8 (0.37) | -0.1 (0.61)
  TPE 6: number analyzed (Participants) | 1 | 1 | 1
  TPE 6 | 4.2 (0) | 3.5 (0) | -0.7 (0)

9. Secondary Outcome: Assessment of Sodium Levels
Description: as for outcome 3
Time Frame: up to 8 days including the 24 hour follow-up
Population: Not all patients received blood draws/multiple TPEs
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Pre-TPE | Post-TPE | Change From Pre-TPE
Number analyzed (Participants) | 41 | 41 | 41
mmol/L
  TPE 1: number analyzed (Participants) | 39 | 36 | 34
  TPE 1 | 140.0 (3.66) | 141.6 (3.23) | 1.6 (2.41)
  TPE 2: number analyzed (Participants) | 24 | 18 | 17
  TPE 2 | 141.2 (3.28) | 142.3 (4.41) | 1.5 (1.84)
  TPE 3: number analyzed (Participants) | 18 | 11 | 11
  TPE 3 | 141.2 (3.87) | 142.9 (5.07) | 1.5 (2.84)
  TPE 4: number analyzed (Participants) | 10 | 8 | 8
  TPE 4 | 140.7 (4.64) | 142.4 (5.13) | 0.8 (1.75)
  TPE 5: number analyzed (Participants) | 6 | 4 | 4
  TPE 5 | 138.8 (3.19) | 141.3 (3.86) | 1.0 (2.16)
  TPE 6: number analyzed (Participants) | 1 | 1 | 1
  TPE 6 | 142.0 (0) | 144.0 (0) | 2.0 (0)

10. Secondary Outcome: Assessment of Leukocyte Levels
Description: as for outcome 3
Time Frame: up to 8 days including the 24 hour follow-up
Population: Not all patients received blood draws/multiple TPEs
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Pre-TPE | Post-TPE | Change From Pre-TPE
Number analyzed (Participants) | 41 | 41 | 41
10^9 cells/L
  TPE 1: number analyzed (Participants) | 41 | 34 | 34
  TPE 1 | 12.8 (6.84) | 13.6 (7.45) | 0.9 (3.80)
  TPE 2: number analyzed (Participants) | 25 | 18 | 18
  TPE 2 | 14.9 (7.45) | 15.3 (6.43) | 1.2 (3.93)
  TPE 3: number analyzed (Participants) | 18 | 9 | 9
  TPE 3 | 13.2 (6.49) | 13.9 (7.20) | -0.5 (2.44)
  TPE 4: number analyzed (Participants) | 9 | 8 | 7
  TPE 4 | 10.8 (6.32) | 12.7 (6.40) | 1.2 (1.14)
  TPE 5: number analyzed (Participants) | 6 | 4 | 4
  TPE 5 | 8.7 (3.17) | 10.7 (3.65) | 1.6 (1.55)
  TPE 6: number analyzed (Participants) | 1 | 1 | 1
  TPE 6 | 3.7 (0) | 7.0 (0) | 3.3 (0)

11. Secondary Outcome: Assessment of Erythrocyte Levels
Description: as for outcome 3
Time Frame: up to 8 days including the 24 hour follow-up
Population: Not all patients received blood draws/multiple TPEs
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | Pre-TPE | Post-TPE | Change From Pre-TPE
Number analyzed (Participants) | 41 | 41 | 41
10^12 cells/L
  TPE 1: number analyzed (Participants) | 41 | 34 | 34
  TPE 1 | 4.0 (0.70) | 4.1 (0.81) | 0.1 (0.26)
  TPE 2: number analyzed (Participants) | 25 | 18 | 18
  TPE 2 | 3.6 (0.60) | 3.7 (0.68) | 0.1 (0.27)
  TPE 3: number analyzed (Participants) | 18 | 9 | 9
  TPE 3 | 3.6 (0.70) | 3.8 (0.60) | 0.1 (0.26)
  TPE 4: number analyzed (Participants) | 9 | 8 | 7
  TPE 4 | 3.7 (0.67) | 3.4 (0.71) | 0.1 (0.17)
  TPE 5: number analyzed (Participants) | 6 | 4 | 4
  TPE 5 | 3.9 (0.96) | 3.2 (0.35) | -0.1 (0.49)
  TPE 6: number analyzed (Participants) | 1 | 1 | 1
  TPE 6 | 2.9 (0) | 2.8 (0) | -0.1 (0)

12. Secondary Outcome: Assessment of Hemoglobin Levels
Description: as for outcome 3
Time Frame: up to 8 days including the 24 hour follow-up
Population: Not all patients received blood draws/multiple TPEs
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Pre-TPE | Post-TPE | Change From Pre-TPE
Number analyzed (Participants) | 41 | 41 | 41
g/dL
  TPE 1: number analyzed (Participants) | 41 | 34 | 34
  TPE 1 | 11.5 (1.94) | 12.1 (2.22) | 0.4 (0.74)
  TPE 2: number analyzed (Participants) | 25 | 18 | 18
  TPE 2 | 10.7 (1.79) | 11.0 (2.03) | 0.3 (0.74)
  TPE 3: number analyzed (Participants) | 18 | 9 | 9
  TPE 3 | 10.4 (1.90) | 11.2 (2.03) | 0.3 (0.70)
  TPE 4: number analyzed (Participants) | 9 | 8 | 7
  TPE 4 | 10.6 (1.61) | 9.9 (1.94) | -0.1 (0.67)
  TPE 5: number analyzed (Participants) | 6 | 4 | 4
  TPE 5 | 10.9 (2.13) | 9.4 (1.06) | -0.5 (1.44)
  TPE 6: number analyzed (Participants) | 1 | 1 | 1
  TPE 6 | 8.7 (0) | 8.3 (0) | -0.4 (0)

13. Secondary Outcome: Assessment of Hematocrit Levels
Description: as for outcome 3
Time Frame: up to 8 days including the 24 hour follow-up
Population: Not all patients received blood draws/multiple TPEs
Measure: Mean (Standard Deviation); unit: % of the blood that is red blood cells
Arm/Group | Pre-TPE | Post-TPE | Change From Pre-TPE
Number analyzed (Participants) | 41 | 41 | 41
% of the blood that is red blood cells
  TPE 1: number analyzed (Participants) | 41 | 34 | 34
  TPE 1 | 34.1 (5.31) | 35.6 (6.44) | 1.1 (2.12)
  TPE 2: number analyzed (Participants) | 25 | 18 | 18
  TPE 2 | 31.7 (4.75) | 32.8 (5.24) | 0.8 (2.39)
  TPE 3: number analyzed (Participants) | 18 | 9 | 9
  TPE 3 | 31.0 (4.98) | 33.3 (5.00) | 1.0 (2.37)
  TPE 4: number analyzed (Participants) | 9 | 8 | 7
  TPE 4 | 31.7 (4.29) | 30.2 (5.50) | 0.6 (1.25)
  TPE 5: number analyzed (Participants) | 6 | 4 | 4
  TPE 5 | 32.9 (5.73) | 28.8 (2.95) | -1.2 (4.03)
  TPE 6: number analyzed (Participants) | 1 | 1 | 1
  TPE 6 | 27.7 (0) | 26.1 (0) | -1.6 (0)

14. Secondary Outcome: Assessment of Mean Corpuscular Volume Levels
Description: as for outcome 3
Time Frame: up to 8 days including the 24 hour follow-up
Population: Not all patients received blood draws/multiple TPEs
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | Pre-TPE | Post-TPE | Change From Pre-TPE
Number analyzed (Participants) | 41 | 41 | 41
fL
  TPE 1: number analyzed (Participants) | 41 | 34 | 34
  TPE 1 | 86.4 (6.96) | 86.8 (6.68) | 0.2 (1.21)
  TPE 2: number analyzed (Participants) | 25 | 18 | 18
  TPE 2 | 88.1 (7.46) | 90.0 (6.91) | 0.3 (1.55)
  TPE 3: number analyzed (Participants) | 18 | 9 | 9
  TPE 3 | 88.2 (11.38) | 87.8 (3.57) | -0.1 (1.55)
  TPE 4: number analyzed (Participants) | 9 | 8 | 7
  TPE 4 | 87.0 (7.90) | 89.9 (6.78) | -0.3 (2.01)
  TPE 5: number analyzed (Participants) | 6 | 4 | 4
  TPE 5 | 85.9 (9.30) | 90.2 (7.02) | -0.1 (2.13)
  TPE 6: number analyzed (Participants) | 1 | 1 | 1
  TPE 6 | 95.0 (0) | 93.0 (0) | -2.0 (0)

15. Secondary Outcome: Assessment of Mean Corpuscular Hemoglobin Levels
Description: as for outcome 3
Time Frame: up to 8 days including the 24 hour follow-up
Population: Not all patients received blood draws/multiple TPEs
Measure: Mean (Standard Deviation); unit: pg
Arm/Group | Pre-TPE | Post-TPE | Change From Pre-TPE
Number analyzed (Participants) | 41 | 41 | 41
pg
  TPE 1: number analyzed (Participants) | 41 | 34 | 34
  TPE 1 | 29.0 (2.54) | 29.4 (2.18) | 0.1 (0.70)
  TPE 2: number analyzed (Participants) | 25 | 18 | 18
  TPE 2 | 29.6 (2.47) | 30.2 (2.48) | 0.1 (0.77)
  TPE 3: number analyzed (Participants) | 18 | 9 | 9
  TPE 3 | 29.2 (2.19) | 29.4 (1.31) | -0.2 (0.58)
  TPE 4: number analyzed (Participants) | 9 | 8 | 7
  TPE 4 | 28.9 (2.41) | 29.2 (1.50) | -0.8 (1.18)
  TPE 5: number analyzed (Participants) | 6 | 4 | 4
  TPE 5 | 28.3 (2.74) | 29.4 (1.75) | -0.4 (0.31)
  TPE 6: number analyzed (Participants) | 1 | 1 | 1
  TPE 6 | 29.8 (0) | 29.6 (0) | -0.2 (0)

16. Secondary Outcome: Assessment of Mean Corpuscular Hemoglobin Concentration Levels
Description: as for outcome 3
Time Frame: up to 8 days including the 24 hour follow-up
Population: Not all patients received blood draws/multiple TPEs
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Pre-TPE | Post-TPE | Change From Pre-TPE
Number analyzed (Participants) | 41 | 41 | 41
g/dL
  TPE 1: number analyzed (Participants) | 41 | 34 | 34
  TPE 1 | 33.6 (1.38) | 33.9 (1.20) | 0.1 (0.75)
  TPE 2: number analyzed (Participants) | 25 | 18 | 18
  TPE 2 | 33.6 (1.35) | 33.6 (1.58) | 0 (0.97)
  TPE 3: number analyzed (Participants) | 18 | 9 | 9
  TPE 3 | 33.4 (2.17) | 33.5 (1.43) | -0.2 (0.91)
  TPE 4: number analyzed (Participants) | 9 | 8 | 7
  TPE 4 | 33.2 (1.16) | 32.6 (1.19) | -0.8 (1.15)
  TPE 5: number analyzed (Participants) | 6 | 4 | 4
  TPE 5 | 33.1 (1.75) | 32.6 (1.21) | -0.5 (0.62)
  TPE 6: number analyzed (Participants) | 1 | 1 | 1
  TPE 6 | 31.4 (0) | 31.8 (0) | 0.4 (0)

17. Secondary Outcome: Assessment of Mean Red Cell Distribution Width Levels
Description: as for outcome 3
Time Frame: up to 8 days including the 24 hour follow-up
Population: Not all patients received blood draws/multiple TPEs
Measure: Mean (Standard Deviation); unit: % red blood cell variation volume/size
Arm/Group | Pre-TPE | Post-TPE | Change From Pre-TPE
Number analyzed (Participants) | 41 | 41 | 41
% red blood cell variation volume/size
  TPE 1: number analyzed (Participants) | 41 | 34 | 34
  TPE 1 | 14.4 (2.66) | 13.9 (1.94) | 0.0 (0.26)
  TPE 2: number analyzed (Participants) | 25 | 18 | 18
  TPE 2 | 14.6 (2.83) | 15.0 (3.02) | 0.1 (0.37)
  TPE 3: number analyzed (Participants) | 18 | 9 | 9
  TPE 3 | 15.2 (3.18) | 15.0 (2.31) | -0.1 (0.33)
  TPE 4: number analyzed (Participants) | 9 | 8 | 7
  TPE 4 | 16.2 (3.10) | 16.5 (3.10) | 0.0 (0.25)
  TPE 5: number analyzed (Participants) | 6 | 4 | 4
  TPE 5 | 17.1 (3.04) | 18.6 (3.24) | 0.3 (0.52)
  TPE 6: number analyzed (Participants) | 1 | 1 | 1
  TPE 6 | 18.2 (0) | 18.0 (0) | -0.2 (0)

18. Secondary Outcome: Assessment of Mean Ionized Calcium Levels
Description: Blood samples compare levels before each TPE (therapeutic plasma exchange), during each TPE, and after each TPE. Pre-TPE is within 24 hours before TPE start; Follow-Up is 24 (+/-2) hours after TPE end.
Time Frame: up to 8 days including the 24 hour follow-up
Population: Not all patients received blood draws/multiple TPEs
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- During TPE: Value during TPE
- Change From Pre-TPE to During TPE: Mean change from Pre-TPE to During TPE
- Follow-Up: Follow-up is 24 (+/-2) hours after TPE end.
- Change From Pre-TPE to Follow-Up: Mean change in level from Pre-TPE to Follow-Up
Arm/Group | Pre-TPE | During TPE | Change From Pre-TPE to During TPE | Follow-Up | Change From Pre-TPE to Follow-Up
Number analyzed (Participants) | 41 | 41 | 41 | 41 | 41
mmol/L
  TPE 1: number analyzed (Participants) | 39 | 38 | 36 | 30 | 28
  TPE 1 | 1.225 (0.0731) | 1.129 (0.1541) | -0.093 (0.1583) | 1.194 (0.0852) | -0.030 (0.0927)
  TPE 2: number analyzed (Participants) | 23 | 23 | 20 | 16 | 14
  TPE 2 | 1.212 (0.0678) | 1.192 (0.1224) | -0.001 (0.0967) | 1.204 (0.0832) | 0.026 (0.1203)
  TPE 3: number analyzed (Participants) | 18 | 15 | 15 | 12 | 12
  TPE 3 | 1.165 (0.2119) | 1.181 (0.1062) | 0.020 (0.1696) | 1.224 (0.0926) | 0.026 (0.0684)
  TPE 4: number analyzed (Participants) | 9 | 10 | 9 | 9 | 8
  TPE 4 | 1.205 (0.0763) | 1.265 (0.1060) | 0.062 (0.0805) | 1.204 (0.0666) | 0.011 (0.0995)
  TPE 5: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
  TPE 5 | 1.200 (0.0452) | 1.240 (0.1039) | 0.040 (0.0640) | 1.168 (0.0948) | -0.032 (0.1089)
  TPE 6: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  TPE 6 | 1.248 (0) | 1.148 (0) | -0.100 (0) | 1.173 (0) | -0.075 (0)

19. Secondary Outcome: Investigator's Assessment of Overall Safety
Description: Excellent: defined as the treatment was well tolerated by the patient; Moderate: defined as Adverse Drug Reaction (ADR(s)) were observed, but easily resolved or not clinically significant; Poor: defined as ADR(s) were observed requiring significant medical intervention
Time Frame: up to 8 days including the 24 hour follow-up
Population: Not all patients received multiple TPEs
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Patients Undergoing TPE
Number analyzed (Participants) | 41
Participants
  Patients Who Underwent TPE 1: Excellent | 37
  Patients Who Underwent TPE 1: Moderate | 4
  Patients Who Underwent TPE 1: Poor | 0
  Patients Who Underwent TPE 2: number analyzed (Participants) | 26
  Patients Who Underwent TPE 2: Excellent | 25
  Patients Who Underwent TPE 2: Moderate | 1
  Patients Who Underwent TPE 2: Poor | 0
  Patients Who Underwent TPE 3: number analyzed (Participants) | 18
  Patients Who Underwent TPE 3: Excellent | 18
  Patients Who Underwent TPE 3: Moderate | 0
  Patients Who Underwent TPE 3: Poor | 0
  Patients Who Underwent TPE 4: number analyzed (Participants) | 10
  Patients Who Underwent TPE 4: Excellent | 9
  Patients Who Underwent TPE 4: Moderate | 1
  Patients Who Underwent TPE 4: Poor | 0
  Patients Who Underwent TPE 5: number analyzed (Participants) | 6
  Patients Who Underwent TPE 5: Excellent | 6
  Patients Who Underwent TPE 5: Moderate | 0
  Patients Who Underwent TPE 5: Poor | 0
  Patients Who Underwent TPE 6: number analyzed (Participants) | 1
  Patients Who Underwent TPE 6: Excellent | 1
  Patients Who Underwent TPE 6: Moderate | 0
  Patients Who Underwent TPE 6: Poor | 0

ADVERSE EVENTS:
Time Frame: Up to 8 days
Description: ADRs will be elicited using a standard non-leading question such as "How have you been since the last evaluation?" If children or adolescent patients are unable to adequately understand and respond to this question, the information will be obtained from the patient's guardian and/or Investigator or study nurse
Arm/Group | Pediatric Patients Undergoing TPE Age Group 1 | Pediatric Patients Undergoing TPE Age Group 2 | Pediatric Patients Undergoing TPE Age Group 3 | All Patients
All-Cause Mortality (participants affected / at risk) | 1/15 | 0/13 | 0/13 | 1/41
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/13 | 0/13 | 1/41
Other Adverse Events (participants affected / at risk) | 0/15 | 3/13 | 1/13 | 4/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pediatric Patients Undergoing TPE Age Group 1 (N=15) | Pediatric Patients Undergoing TPE Age Group 2 (N=13) | Pediatric Patients Undergoing TPE Age Group 3 (N=13) | All Patients (N=41)
Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pediatric Patients Undergoing TPE Age Group 1 (N=15) | Pediatric Patients Undergoing TPE Age Group 2 (N=13) | Pediatric Patients Undergoing TPE Age Group 3 (N=13) | All Patients (N=41)
Citrate toxicity (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Inflammatory marker increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-10-19): https://cdn.clinicaltrials.gov/large-docs/78/NCT01938378/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-22): https://cdn.clinicaltrials.gov/large-docs/78/NCT01938378/SAP_001.pdf